CLINICAL TRIAL: NCT03981757
Title: Study of Regional Cerebral Oxygenation and Brain Blood Volume Changes During Carotid Endarterectomy Using the NeurOS System
Acronym: COBBV-CE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor withdrew
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Jiapeng Huang, Principal Investigator, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19.0273
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Carotid Disease
Keywords: carotid surgery; cerebral oxygenation; brain blood volume

STUDY DESIGN:
Intervention Model Description: Patients will have NeurOS pads placed on their foreheads. Continuous monitoring of arterial blood pressure, cerebral oxygenation and brain blood volume index for the whole length of surgery will be recorded and saved in a USB drive for retrieval and analysis. Key point data include: Baseline, Anesthesia Induction, Incision, Carotid Clamping, Clamp Release and Skin Closure. These key points data will be extracted for analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NeurOS Group (Experimental): Apply the single use NeurOS cerebral oximetry sensor adhesive onto patients' head who are going to have CEA surgery in the operating room before anesthesia induction.
  Interventions: Device: NeurOS

INTERVENTIONS:
Device: NeurOS — NeurOS system pads will be placed on patients' head for monitoring.

SUMMARY:
Study of Regional cerebral Oxygenation and Brain Blood Volume changes during Carotid Endarterectomy using the NeurOS system

DETAILED DESCRIPTION:
1. Title of the Research Project： Study of Regional cerebral Oxygenation and Brain Blood Volume change during Carotid Endarterectomy using the NeurOS system (COBBV-CE Trial)
2. Background/Problem Statement: The use of regional cerebral oxygenation (rSO2) monitoring has grown clinically, even becoming the standard of care in some institutions. Monitoring of intracranial tissue oxygenation is fundamentally possible because light in the near infrared spectrum (700-900nm) penetrates bone, muscle, and other tissue. Oxyhemoglobin and deoxyhemoglobin have distinct peak absorption spectra, but there is an isobestic wavelength (i.e., wavelength for which the peak absorption of light is similar for oxyhemoglobin and deoxyhemoglobin, approximately 810nm) for absorption by total hemoglobin. Determination of rScO2 thus is possible with transmission of just 2 wavelengths of near-infrared spectroscopy (NIRS) to determine the relative concentrations of oxyhemoglobin versus total hemoglobin. A decrease in rSO2 from baseline >20% or an absolute rSO2 value <50% often is reported in clinical investigation as representing a clinically meaningful reduction or "desaturation."

Cerebral autoregulation was found to be impaired in carotid stenosis patients. Recent research found that NIRS allows continuous non-invasive monitoring of cerebral oxygenation during CEA, with high sensitivity and acceptable specificity in predicting cerebral ischemia and the need for shunting, which makes it an attractive alternative to stump pressure. Regional cerebral oxygenation provides a clinically acceptable surrogate of cerebral blood flow (CBF) for clinical autoregulation monitoring. Monitoring CBF autoregulation with rSO2 has many clinically attractive features, including the following: It is noninvasive, monitoring requires little caregiver intervention, and it has sufficient resolution to discriminate the lower autoregulatory threshold to prevent brain ischemia. On the other hand, simply raising mean blood pressure targets, however, may not necessarily be beneficial because for some individuals this may result in blood pressure above the upper limit of autoregulation, which potentially could lead to cerebral hyperperfusion, increasing cerebral embolic load and/or enhancing cerebral edema in the setting of systemic inflammatory response to cardiac surgery. Individualizing blood pressure during CPB based on physiological endpoints such as rSO2 monitoring, rather than empiric targets, may provide a means for modifying the risk for renal injury and major organ morbidity and possibly mortality. In patients undergoing combined CEA and CABG surgery, it was found that the utility of NIRS could compliment patient selection for CEA as well as for individual patient management during. The brain blood volume changes during CEA has not been defined and would be significantly reduced by carotid artery clamping during CEA. Abnormalities of the circle of Willis would contribute to reduced brain blood volume. The combination of rSO2 and cerebral blood volume would be very helpful to prevent mal-perfusion of either side of the brain. Postoperative delirium could happen after CEA due to reperfusion of the previously ischemic regions of the brain, regulation of cerebral blood volume after CEA would also prove beneficial to prevent postoperative delirium.

Problem Statement: Disposable rSO2 sensors are costly and is becoming a rate limiting factor hindering its widespread clinical use. Reusable sensors like NeurOS cerebral oximetry are only a fraction of cost with similar performances in healthy volunteers. We will use NeurOS in accordance with its approved labeling and indications by FDA. CEA surgery has significant variations and great clinical importance of cerebral oxygenation during different stages of surgery. Blood volume changes before, during and after CEA have not been studied previously and could provide critical information to prevent postoperative cognitive changes. The NeurOS system calculates the sum of attenuation of two wavelengths to provide brain blood volume index (BVI) continuously.

Patients presenting for carotid endarterectomy face two challenges during surgery. First, how to protect the brain when the carotid artery is clamped, meaning no blood flow to that side of the brain from this carotid artery. Second, how to prevent hyperemia when the carotid artery is open and might provide too much blood flow to the brain. Our aim is to study the cerebral oxygenation and brain blood volume changes during carotid endarterectomy and identify whether they are related to clinical outcomes.

3. Objectives:

1. To study the cerebral oxygenation changes with NeurOS system and correlate desaturation with outcomes.
2. To study the brain blood volume changes during CEA surgery and correlate with clinical outcomes.

4. Study Design/Methodology: Patients will have NeurOS pads placed on their foreheads. Continuous monitoring of arterial blood pressure, cerebral oxygenation and brain blood volume index for the whole length of surgery will be recorded and saved in a USB drive for retrieval and analysis. Key point data include: Baseline, Anesthesia Induction, Incision, Carotid Clamping, Clamp Release and Skin Closure. These key points data will be extracted for analysis.

1. . Sample selection and size: 100 consecutive carotid endarterectomy patients at Jewish Hospital, Louisville, KY (6 months to recruit)
2. . Describe the proposed intervention: Apply the single use NeurOS cerebral oximetry sensor adhesive onto patients' forehead who are going to have CEA surgery in the operating room before anesthesia induction.
3. . Data collection procedures, instruments used, and methods for data quality control: Anesthesia providers (attending anesthesiologists, residents and CRNAs) provide routine anesthesia care for CEA surgery. NeurOS rSO2 reading are automatically recorded in the VO200-NeurOS Cerebral Oximetry Monitor and the INOVS Monitor respectively. Significant events (Baseline, Anesthesia Induction, Incision, Carotid Clamping, Clamp Release and Skin Closure) will be marked manually by the anesthesia providers in the NeurOS system. Brain blood volume index will be automatically recorded and retracted from the NeurOS system once surgery is over. All data will be downloaded from the system into an encrypted USB drive for storage and analysis. Data quality control will be ensured by the individual system alarms for poor signals and be corrected by anesthesia providers.
4. . Unit of analysis and observation: Cerebral Oxygenation in percentage of oxyhemoglobin. Brain blood volume index in the sum of attenuation of two wavelengths.

5. Subject Recruitment Methods: All patients presenting to Jewish Hospital for CEA surgery will be contacted for potential recruitment on the day of surgery in the preoperative area.

6. Informed Consent Process/Complete Waiver Process: Informed consent will be provided to all participants.

7. Research Procedures:

In all consented patients, baseline cerebral oxygenation and brain blood volume index will be obtained at room air or baseline oxygen requirement level in the NeurOS systems. Both NeurOS rSO2 and brain blood volume indexes will be continuously recorded and saved in the respective system throughout the whole CEA surgery. General anesthesia will be induced by using O2 administered via face mask and IV fentanyl 1μg/ kg, propofol 2-3mg/kg and rocuronium 1mg/kg. Maintenance of anesthesia was achieved with inhaled isoflurane in air/oxygen mixture and muscle relaxation using intermittent boluses of rocuronium. Fentanyl will be used as supplemental analgesia. Normocapnic ventilation was maintained. Upon completion of surgery, titrated doses of protamine will be administered to reverse the anticoagulant action of heparin, targeting to achieve baseline preoperative Activated clotting Time.

After the surgery, all rSO2 and brain blood volume index data are downloaded into an encrypted USB drive for analysis and storage.

8. Minimizing Risks:

1. All HIPPA related information will be stored in a private computer in a password protected computer.
2. Cleaning of cables, monitors and reusable equipment are performed after each use.
3. Standard electrical precautions will be followed to prevent electrical shock to providers and patients.

9. Plan for Analysis of Results:

* Trend graphs of NeurOS brain blood volume index, arterial blood pressure and cerebral oxygenation will be plotted together to identify correlations among them.
* Cerebral oxygenation and brain blood volume index deviation from the baseline at each key point will be analyzed to identify whether these critical moments affect cerebral oxygenation and the brain blood volume. Clinical outcomes data will be collected on 30-day mortality and strokes to identify whether abnormal cerebral oxygenation and brain blood volume directly (too high or too low, Area Under or Above the Curve) affects clinical outcomes.
* Programs to be used for data analysis: Software R

  10. Research Materials, Records, and Privacy: Identify the sources of research material obtained from individually identifiable living human subjects: Prospective noninvasive data on cerebral oxygenation and brain blood volume during cardiac surgery. Please see data collection form.

Indicate what information (records, data, etc.) will be recorded and whether use will be made of existing records or data: Cerebral oxygenation and brain blood volume. They will be recorded in the medical charts.

Explain why this information is needed to conduct the study: These data are necessary to identify outcomes for these patients.

Specify how the data will be de-identified (if applicable), who has access to the data, where the data will be stored and how the researcher will protect both the data with respect to privacy and confidentiality. Address physical security measures (e.g., locked facility, limited access); data security (e.g., password-protection, data encryption); safeguards to protect identifiable research information (e.g., coding or links): Once required information is collected, HIPPA information will be deleted. All HIPPA related information will be stored in a private computer in a password protected computer. No links will be provided to the public.

ELIGIBILITY:
Inclusion Criteria:

Having carotid endarterectomy at Jewish Hospital, Louisville, KY Agree to study protocol No allergy to either INOVS or NeurOS system pads

Exclusion Criteria:

Refusal to participate Emergency surgery Allergy to either INOVS or NeurOS system pads

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Regional Cerebral Oxygenation | From the beginning of surgery until the end of surgery for each patient enrolled
  Regional Cerebral Oxygenation during Carotid Endarterectomy

SECONDARY OUTCOMES:
NeurOS Brain Blood Volume | From the beginning of surgery until the end of surgery for each patient enrolled
  NeurOS Brain Blood Volume during Carotid Endarterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Jiapeng Huang, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No